CLINICAL TRIAL: NCT01098734
Title: A 12-week Efficacy Evaluation of WBI-1001 Cream in Patients With Atopic Dermatitis: A Multi-centered, Double-blinded Study (6-week Placebo-controlled Phase Followed by a 6-week Non-placebo Controlled Phase).
Brief Title: Non-steroid, Atopic Dermatitis Phase IIb 12-week Trial; Topical WBI-1001 Cream
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Welichem Biotech Inc. (Industry)
Responsible Party: R. Bissonnette, MD, MSc, FRCPC, Innovaderm Research Inc.
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: WBI-1001-202 : # 133148; # 133148 (Registry Identifier: Health Canada: Therapeutic Products Directorate)
Record Dates: First submitted 2010-04-01; First posted 2010-04-05 (Estimated); Last update posted 2011-06-13 (Estimated); Status verified 2011-06

CONDITIONS: Dermatitis, Atopic
Keywords: non-steroid; anti-inflammatory; skin disease; topical cream; small molecule; atopic dermatitis; eczema
MeSH Terms: conditions — Dermatitis, Atopic; Skin Diseases; Eczema | interventions — tapinarof

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Placebo Comparator): 0%; vehicle cream
  Interventions: Drug: WBI-1001
- Group 2 (Active Comparator): 0.5% WBI-1001 cream
  Interventions: Drug: WBI-1001
- Group 3 (Active Comparator): 1.0% WBI-1001 cream
  Interventions: Drug: WBI-1001

INTERVENTIONS:
Drug: WBI-1001 — A 12-week study to assess the efficacy, safety and tolerability of topically applied WBI-1001 creams. First 6 weeks will be double-blinded, placebo-controlled and the following 6 weeks will be double-blinded, non-placebo- controlled. After 6 weeks patients in Groups 2 and 3 will continue double-blinded treatment for a further 6 weeks, but patients in Group 1 will enter a 6-week double-blinded phase with one of the two active creams (half treated with 0.5% and half with 1.0% WBI-1001 cream). All patients treated twice daily (BID).

SUMMARY:
Welichem Biotech has developed a small molecule drug candidate, WBI-1001, that selectively targets the pathogenic features of inflammatory skin diseases, including atopic dermatitis (a form of eczema).The purpose of this clinical trial is to further test the safety and efficacy of WBI-1001 as a topically applied cream over an extended period of 12 weeks on patients with mild to moderate atopic dermatitis.

DETAILED DESCRIPTION:
A multi-centered, double-blinded Phase IIb study to evaluate the safety and efficacy of the non-steroid, anti-inflammatory WBI-1001 cream in the topical treatment of patients with mild to moderate atopic dermatitis, expressed as lesions up to 20% BSA. For the first 6 weeks patients will be randomized to one of three treatment groups simultaneously in a ratio of 1:1:1.

Group 1: vehicle cream (placebo), BID; Group 2: 0.5% WBI-1001 cream, BID; Group 3:1.0% WBI-1001 cream, BID. Patients randomized to treat all lesion areas.

After the first 6 weeks all patients will be treated, non-placebo controlled, with WBI-1001 cream. The Group 1 patients will enter a double-blinded phase for a further 6 weeks with half of them being treated BID with 0.5% and half with 1.0% WBI-1001 cream. Groups 2 and 3 will continue with their treatments unchanged for the remaining 6 weeks.

During the treatment period, patients will apply the cream (BID) from the kit that they have been provided, and they will visit the study centre at prescribed times for assessment of efficacy, safety and tolerability. After completion of the 12-week treatment period patients will have a 2-week follow-up visit.

Patients who withdraw from the study before Day 42 for reasons other than a treatment related AE will be replaced so that at least 40 patients per group will complete the placebo-controlled phase.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic atopic dermatitis (Hanifin's criteria) for greater than 6 months with a minimum of 5% and a maximum of 20% BSA.
* IGA scores of 2-4 at Day 0.
* WOCBP must have a negative serum beta-hCG pregnancy test before randomization, and they and their male partners must take pregnancy precautions for the duration of the study, as also must male patients.
* Willing to comply with Protocol and attend all visits.
* Provide written informed consent prior to entering study procedures.
* Patient has no latent or active tuberculosis infection according to medical history or current examination and tests.

Exclusion Criteria:

* Pregnancy or lactation.
* Spontaneously improving or rapidly deteriorating atopic dermatitis.
* Presence of atopic dermatitis on only hands and/or feet.
* Any skin disease other than atopic dermatitis that might interfere with clinical assessment or put patient at risk.
* Active allergic contact dermatitis or other non-atopic forms of atopic dermatitis.
* Other concommitant serious illness or medical condition, virus or renal insufficiency, or clinically significant abnormality that could put patient at risk during the study.
* History of neurological/psychiatric disorders including psychotic disorders, dementia or any other reason that would interfere with the patient's participation.
* Systemic immunomodulatory therapies for other conditions within 4 weeks prior to the baseline visit.
* Any phototherapy, photochemotherapy or systemic atopic dermatitis therapy within 2 weeks of the baseline visit.
* Prolonged exposure to natural or artificial sources of UV within 4 weeks prior to baseline visit or intention to have such exposure during the study.
* Topical atopic dermatitis therapies (including corticosteroids and calcineurins) in the areas to be treated within 2 weeks prior to baseline.
* Alcohol abuse in the last 2 years.
* Allergic history to any of the non-medical ingredients of the study cream.
* Treatment with an investigational drug within one month of Day 0 or current participation in another clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2009-11; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Investigator's Global Assessment (IGA) score | The change from baseline to 6 weeks.
  To evaluate the efficacy of the 0.5% and 1.0% WBI-1001 creams in comparison with the vehicle placebo.

SECONDARY OUTCOMES:
Eczema Area and Severity Index (EASI) score | The change from baseline to 6 weeks.
  Comparison over time with the placebo.
Scoring Atopic Dermatitis (SCORAD) Index. | Change from baseline to 6 weeks.
  Comparison over time with the placebo.
Clinical laboratory tests (haematology, urine) and vital signs. | From baseline through 12 weeks+2 weeks follow-up
Adverse events | From baseline through 12 weeks+2 weeks follow-up
BSA and pruritus. | From baseline through 6 weeks.
  Comparison over time with placebo.
Longterm change in IGA score of WBI-1001 cream groups. | Change from baseline through 12 weeks
  Long term comparison, non-placebo, of the 0.5% and 1.0% cream treated groups of patients
Statistically significant improvement in the rate of "Treatment Success" with 0.5% and 1.0% WBI-1001 creams compared with placebo. | First 6 weeks
  "Treatment Success" is defined as a patient who (1) achieves "clear" (IGA=0) or "almost clear" (IGA=1) on a five-point IGA scale or (2) has a minimum of 2-point improvement in IGA score over the baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Liren Tang, Ph.D, Study Director — Sponsor GmbH
Locations (5):
- Canada (5):
  - Guilford Dermatology Associates, Surrey, British Columbia
  - Department of Dermatology and Skin Sciences, UBC, Vancouver, British Columbia
  - Windsor Clinical Research Inc., Windsor, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
  - Centre de Recherche Dermatologique du Quebec, Québec, Quebec